CLINICAL TRIAL: NCT05673538
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TT-00973-MS Tablets in Patients With Advanced Solid Tumors
Brief Title: TT-00973-MS Tablets in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT00973CN02
Record Dates: First submitted 2022-11-03; First posted 2023-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TT-00973-MS Tablets (Experimental): TT-00973-MS tablets will be administered at the starting dose of 2mg. Subsequently, patients will be enrolled according to the standard 3+3 dose escalation design.
  Interventions: Drug: TT-00973-MS tablets treatment

INTERVENTIONS:
Drug: TT-00973-MS tablets treatment — The dose levels to be tested in the dose escalation cohorts are 2, 5, 10, 17, 25, 32, 40 and 50mg QD. All the subjects will receive TT-00973-MS tablets QD until disease progression or occurrence of intolerant adverse reactions.

SUMMARY:
This study is a multicenter, open-label, phase 1 study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of TT-00973-MS tablets in patients with solid tumors.

DETAILED DESCRIPTION:
A modified 3+3 design will be used to determine the maximum tolerated dose(MTD) during dose escalation period. Futher expansion period will enroll additional 12~18 patients at the appropriate dose to futher evaluate the safety and preliminary efficacy of TT-00973-MS.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Histologically or cytologically confirmed advanced malignant solid tumors, eligible patients have failed standard treatment, have no standard treatment, or are not suitable for standard treatment at this stage as determined by the investigator.
3. Must have at least one evaluable lesion in dose escalation period and one unidimensional measurable lesion according to RECIST version 1.1;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Life expectancy ≥3 months;
6. Patients must have adequate organ functions as indicated by the following screening laboratory values: ANC ≥ 1.5×10^9/L; PLT ≥ 75×10^9/L; Hb ≥ 90 g/L; TBIL ≤ 1.5×ULN；ALT和AST ≤ 3×ULN(ALT and AST≤5×ULN for subjects with liver cancer or hepatic metastases); Cr ≤ 1.5×ULN or CLcr >50mL/min(according to Cockcroft-Gault); APTT≤ 1.5×ULN; INR≤ 1.5×ULN.
7. Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose, and female subjects of childbearing potential have a negative pregnancy test at baseline.
8. Written, signed, and dated informed consent to participate in this study.

Exclusion Criteria:

1. Previous treatment with any AXL inhibitors.
2. Anticancer treatment including radiation therapy, chemotherapy, hormonal therapy, molecular targeted therapy, or immunotherapy within 4 weeks prior to the first dose of TT-00973-MS.
3. Have systematic hormonal therapy(prednisone>10mg/d or similar drugs with equivalent dose)or immunosuppressor therapy with 14 days prior to the first dose of study drug, except using topical,ocular,intra-articular,intranasal,inhaled corticosteroids,and preventive therapy using corticosteroids in short period(for instance,to prevent hypersensitivity to contrast media).
4. Participate in other clinical trials within 4 weeks prior to first dose administration.
5. Concomitant use of any strong inhibitors or inducers of CYP3A4, and can not withdrawal at least 1 week before the first dose of study drug.
6. History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
7. Adverse events occurred during previous anticancer therapy have not been recovered to ≤1(CTCAE 5.0)except toxicity with no significant risk determined by investigators such as alopecia.
8. Evidence of central nervous system (CNS) metastases accompanied with clinical symptoms, or other evidence of uncontrolled CNS metastases judged by investigators that the patient should not participate in the study.
9. Presence of grade 3 or 4 gastrointestinal bleeding or esophageal and gastric varices in three months prior to enrollment.
10. Have moderate or severe cardiac disease, including but not limited to severe arrhythmias or abnormal cardiac conduction, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block,QTcF≥450 ms for male, QTcF≥470 ms for female, or other structural heart disease with high risk as determined by investigators;history of acute coronary syndrome, congestive heart failure,aortic dissection,stroke or other≥grade 3 cardiovascular and cerebrovascular events within 6 months prior to the first dose of study drug;New York Heart Association (NYHA) Class II or greater heart failure, or LVEF<50% ;uncontrolled hypertension;any risk factors to increase QTc or arrhythmias, including heart failure,hypokalemia,congenital long QTc syndrome,family history of long QT interval syndrome or history of unexplained sudden death occurred in first degree relative less than 40 years of age, or using any concomitant medication known to produce QTc prolongation.
11. Have active infection requiring systemic with one week prior to the first dose the study drug.
12. Infection with hepatitis B virus(HBV DNA≥10^3 copies/mL )and hepatitis C virus(HCV RNA above the lower limit of detection) .
13. History of immune deficiency including HIV antibody positive.
14. Have received any live or attenuated live vaccine within 4 weeks prior to the first dose.
15. Major surgery(not include biopsy),or significant traumatism,or requiring selective operation within 4 weeks prior to study entry.
16. Inability to swallow the drug, or severe gastrointestinal disease affecting absorption of the drug.
17. Uncontrolled effusion in the third space, not suitable for entry as determined by the investigator.
18. With alcohol or drug abuse disorder.
19. With mental disorders or non-compliance.
20. Women who are pregnancy or breastfeeding.
21. Judgment by the investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | At the end Cycle 1(each cycle is 28 days)
  To evaluate the incidence of DLT and determine the maximum tolerated dose.
Incidence of adverse events and sevious adverse events | Adverse events are collected from the patient's first dose of TT-00973-MS until 28 days following the last dose of study drug.
  To evaluate the safety and tolerability of TT-00973-MS tablets administered orally in patients with advanced solid tumors. NCI CTCAE 5.0 grading system will be used to determine the severity.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 single dose; pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 28 of Cycle 1
Area under the plasma concentration versus time curve (AUC) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 single dose; pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 28 of Cycle 1
Time to reach maximum plasma concentration (Tmax) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 single dose;pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 28 of Cycle 1
terminal half-life (T1/2) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 single dose;pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 28 of Cycle 1
Objective response rate(ORR) | Up to approximately 1 year
  ORR is defined as the rate of CR and PR.
Objective response rate(DCR) | Up to approximately 1 year
  DCR is defined as the rate of CR, PR and SD.
Progression-free survival(PFS) | Until the date of documented confirmed relapse/progression or death, whichever occurs first, assessed up to 1 year.
  PFS will be calculated from the date of first dose to the date of documented confirmed relapse/progression or death, whichever occurs first.
Duration of response(DOR) | Up to approximately 1 year
  DOR will be calculated as the date of the first documented CR/PR to the date of the first documented confirmed relapse or death, whichever occurs first.
Overall survival(OS) | Up to approximately 1 year
  Overall survival is defined as the time from first dose to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, Principal Investigator — Hunan Cancer Hospital; Nong Yang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (3):
- China (3):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Hunan Cancer Hospital, Changsha, Hunan